CLINICAL TRIAL: NCT05781763
Title: High-intensity Exercise Based on Self-management With Digital Coaching in Patients With Spondyloarthritis: a Randomized Controlled Trial
Brief Title: High-intensity Training in Patients With Spondyloarthritis: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halmstad University (Other)
Responsible Party: Principal Investigator, Emma Haglund, Associate professor in biomedicine, Halmstad University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 350974
Record Dates: First submitted 2023-02-05; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into intervention- and control groups. Simple randomization will be used for equal group allocation at three different rheumatology clinics in southern Sweden. The patients will choose a sealed note in which one of the words "intervention" or "control" is written, when the baseline assessment is completed at the first measurement occasion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT-intervention group (Experimental): 12 weeks of structured high intensity interval training followed by 9 month of self-selected training
  Interventions: Behavioral: High intensity interval training (HIIT)
- Control group (Active Comparator): Continuing with their usual exercise habits during 12 months
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: High intensity interval training (HIIT) — 2 HIIT sessions/week in self-selected activity and type of interval-session with in total 15 minutes interval time (85-90% of MHR) with active rest (50-70% of MHR) between intervals for 12 weeks
  1 self-selected session at moderate or high-intensity/week for 12 weeks Standardized physical and digital coaching by a physiotherapist
  Arms: HIIT-intervention group
Other: Control group — Continuing with exercise as usual during 12 months
  Arms: Control group

SUMMARY:
Project summary

Background: For people diagnosed with a spondyloarthritis (SpA) e.g. ankylosing spondylitis or undifferentiated spondyloarthritis, physical activity and exercise are important components in the self-management. Exercise, in addition to physical and mental symptoms related to the disease can easily feel overwhelming to exercise, and low adherence may result. By studying the effects of high-intensity interval training (HIIT) in comparison with training as usual on physiological, inflammatory, and self-reported disease parameters in patients with SpA, we intend to further investigate the short-term and longitudinal training effects, and refine the knowledge to tailor, coach, and stimulate to self-performed HIIT.

Objective: The purpose of this study is to investigate the short- and long-term effects of high- intensity interval training (HIIT) on physiological, inflammatory, and self-reported health parameters in patients with SpA. The aim is also to study the adherence to physical activity and exercise recommendations.

Design: A randomized controlled trial (RCT) design. Participants: One hundred adults with a confirmed axial SpA from rheumatology clinics in southern Sweden will be recruited and randomized into two groups, the intervention group and the control group.

Intervention: Three high-intensity training sessions per week for three months, of which two interval sessions, with coaching both from a clinical physiotherapist and digital devices (watch and app) followed by nine months with sporadic coaching. The control group will go on with exercise as usual.

Primary outcome: Self-reported disease activity, inflammatory biomarkers (acute phase proteins).

Secondary outcomes: Physical fitness (aerobic capacity (VO2max), blood pressure, grep strength), body composition and self-reported physical function, health status, well-being, pain, fatigue, adherence to physical activity and exercise recommendations, and confidence in one's own ability to manage pain, symptoms and high-intensity exercise, and additional serum biomarkers.

DETAILED DESCRIPTION:
Introduction SpA is an umbrella term for a group of inflammatory diseases with a prevalence that varies between 0.2% - 1.6% globally. SpA can be divided into two forms; axial SpA characterized by inflammation in the spine and pelvic joints, and in peripheral SpA characterized by inflammation in peripheral joints, entesites and dactylites. Recommended treatment consists of a combination of pharmacological and non-pharmacological interventions. The non-pharmacological treatment includes physiotherapy with disease counselling and specific training. There is an increased risk of comorbidity such as cardiovascular disease, obesity, depression and osteoporosis in patients with axSpA. The risk of several of the comorbidities that occur is considered to be reduced through an increased degree of physical activity. The increased cardiovascular risk is considered multifactorial but is partly explained by the chronic systemic inflammation and a low level of physical activity.

The effects of high-intensity interval training (HIIT) with respect to inflammatory biomarkers are poorly studied in individuals with rheumatic diseases. Also, proteins secreted by muscle cells during physical activity, myokines, and their suggested effect to counteract the inflammatory process, need to be further studied. HIIT is believed to be able to affect both the disease outcome and the increased risk of cardiovascular morbidity, but more studies are needed to obtain sufficient evidence along with new biomarkers recently found to affect inflammation that can be implemented in a general maintenance of the individuals' systemic inflammatory status. In the general population, the greatest positive effect is seen on cardiovascular disease and its risk factors during cardio training at a higher intensity. Studies show that individuals with SpA can exercise at a higher intensity level without exacerbating disease activity and that HIIT can reduce inflammation and reduce the cardiovascular risk factors for individuals with SpA.

Despite the overwhelming evidence that exercise will help in the disease management, individuals with the disease still find it difficult to make exercise a sustainable routine in their lives. Previous studies have shown that when a coach-led intervention ends, it is common with a large drop-out rate and that compliance decreases. Changing a behavior should take place gradually and over a long period of time to have the best conditions to become permanent. A person-centered approach with the opportunity to choose activity, and be able to vary activity and training sessions have proven to be important factors that increase compliance with HIIT. Active coaching, registration of heart rate level during training and estimation of perceived effort have all been shown to be important to achieve the right training intensity. Telehealth, in which health coaching is provided via telecommunications and other virtual communication devises outside traditional health care, is considered an important part of modern care, among other things, to encourage change. However, the effects of this type of intervention are still incompletely studied.

The effects of HIIT on physical, inflammatory, and self-reported health parameters needs to be further studied. The knowledge is also scarce on how to tailor the high-intensity training as a part of the self-management for individuals with SpA, with the aim to maintain regular exercise routines and sustainable health over time.

Objectives The purpose of this study is to investigate the short- and long-term effects of self-performed high-intensity interval training (HIIT) on physiological, inflammatory, and self-reported health parameters in patients with SpA. The aim is also to study the adherence to the physical activity and exercise recommendations.

The primary hypothesis in this study is that there will be significant differences between the intervention group and the control group concerning self-reported disease activity, in some of the inflammatory biomarkers (acute phase proteins and pro-inflammatory cytokines), and in adherence to vigorous intensity performed physical activity and exercise both in the short and long term.

The secondary hypothesis is that there will be significant differences between patients in the intervention group and the control group regarding physiological health (aerobic capacity, blood pressure, grip strength, body composition), and self-reported health (physical function, health status, well-being, pain, fatigue, inactivity), and in the confidence in one's own ability to manage pain, symptoms, and high-intensity training, after both three- and twelve-months follow-ups.

Methodology The results of a three-months intervention with high-intensity training, followed by nine months with customized coaching where the intervention group will be motivated and strengthened in their own confidence to continue training regularly at high-intensity levels, will be compared to the control group for primary- and secondary outcomes. The control group continues with their regular physical activity and exercise routines as before.

The patients will be recruited from rheumatological clinics in southern Sweden, through invitation via personal contact by the physiotherapist at the clinic. Participants will be randomly assigned into intervention- and control groups after baseline assessments.The baseline tests include both patients in the experimental and control groups. Baseline tests will include physiological tests, body composition, blood tests, self-reported questionnaire including different health variables, collected during one visit. After 12 weeks of intervention, and after one year the same assessment will be made.

A clinical physiotherapist at each centre will identify eligible patients and, checking the inclusion criteria in the medical record, and screen for cardiovascular or other comorbidities contraindicated for high-intensity training. After showing interest in participating, they will receive oral and written information. An informed consent will be signed by all included patients before the data collection will start. At the initial visit the physiotherapist will start by measuring the chest thumb electrocardiography (ECG). In the event of two repeated deviating results regarding the ECG, the patients will be referred to the health centre for further investigation before any inclusion.

Intervention The patients in the intervention group will be instructed to perform two HIIT/week and one further training session at moderate or high-intensity of their own choice every week mostly on their own for 12 weeks. Structured coaching will be given with support of text messages and a heart rate (HR) feedback from a fitness watch (Polar Ignite, Polar Electro Oy, Kempele, Finland). The approach is based on a person-centered care approach with self-selected activity that engages large muscle groups, such as cycling, Nordic walking, running, swimming, rowing, cross-training. During the first 12 weeks, coach-led sessions are offered on at least three occasions, during week 1, 2 and 7 with the aim of guiding the patients to the right intensity. The intensity will be individually based on the patient's max heart rate (MHR). If necessary, additional coach-led sessions will be offered. After the 12 initial weeks, the intervention continues for another nine months with customized coaching where the patients will be motivated and strengthen in their own confidence to continue with HIIT sessions. During this time, the participants will go on and register the training sessions with the fitness watch, and they will be contacted once a month by their coach for guidance.

The intervention begins with a coach-led interval session during week 1 consisting of 4x4 min intervals with 3 minutes active rest (at 50-70% of MHR) between each interval. The first session will be performed on a stationary bicycle. The session will start with a warm-up to a heart rate of 60-70% of MHR, afterwards the load will be increased to 85% of MHR in the interval with the intention to reach 90% at some point during each interval. Perceived exertion will be assessed with the RPE scale and the goal is to reach at least RPE 17 during the intervals. The session will end with a cool down at <60% MHR. The patient will be able to choose between different interval sessions, but the total time for the intervals in each session should be 15 minutes. In addition to the two HIIT session, the patient will be instructed to perform one further high-intensity training each week at a HR of at least 75% of MHR or at RPE 14. At least one rest day should be planned in between each session.

The continuous monitoring of HR and individual coaching will be based on data available through the fitness watch and a web-based coaching platform. The coaching physiotherapist will log in as a coach and be able to follow the training sessions digitally every week. During the first four weeks, the patients will be contacted once a week by phone. After week 4, the follow-up of each patient will be based on their own wishes, but at least once/month. Three text messages/week will be sent to the patients in the intervention group during the initial 12 weeks with a reminder to stay active.

Data analysis Data analysis will be performed using Microsoft Excel and IBM SPSS (IBM SPSS Statistics for Windows). The level of significance is set to p<0.05. Depending on if the data is normally distributed or not, appropriate statistical method will be used. If normally distributed, the main outcomes will be analyzed with two-way ANOVA. To find a minimum difference between the groups according to self-reported disease activity, a sample size calculation of 50 patients for two subgroups, approximately 100 participants, will be needed to obtain a power of 80% at a significance level of 5%.

Ethics The study will be accomplished in the terms of the Declaration of Helsinki. The Swedish Ethical Review Authority approved the study (2019-04155, 2022-03114-02). All collected study-specific data will be managed confidential and the patients' personal data will be replaced by codes. The results from the routine blood samples will be entered into the medical record in accordance guidelines and the Patient Data Act and data will then retrieved from there. Only researchers in the project will have access to the coded data for the analysis and the results will be presented at group levels. After the analyses are finished the collected data will be stored on a security-protected server at Halmstad University, and the blood samples will be stored in a biobank at FoU Spenshult.

ELIGIBILITY:
Inclusion Criteria:

* Axial SpA (ICD10 diagnosis of M45, M46.0, M46.1, M46.8 and M46.9).
* Fulfilling recommendations for physical activity

Exclusion Criteria:

* Changed TNF and anti-inflammatory medication the previous three months
* Cardiovascular disease
* Comorbidities making high-intensity training inappropriate
* Performing high-intensity interval training on a regular basis

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported disease activity BASDAI | after 3 months
  The disease-specific Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) based on six questions on fatigue, pain, tenderness, and morning stiffness measured with numeric questions (range 0-10). The final score is estimated by calculating the mean score 0-10 (best-worse)
Self-reported disease activity BASDAI | after 12 months
  The disease-specific Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) based on six questions on fatigue, pain, tenderness, and morning stiffness measured with numeric questions (range 0-10). The final score is estimated by calculating the mean score 0-10 (best-worse)
Self-reported disease activity ASDAS-CRP | after 3 months
  Ankylosing Spondylitis Disease Activity Score with C-reactive protein (ASDAS-CRP). Consists of four questions on pain in neck, back, and hip, morning stiffness, well-being, and pain/stiffness in other joints in addition to blood test of CRP. Score 0-4 (<1.3 inactive disease, >3,5 very high disease activity). Equation ASDAS-CRP = 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1)
Self-reported disease activity ASDAS-CRP | after 12 months
  Ankylosing Spondylitis Disease Activity Score with C-reactive protein (ASDAS-CRP). Consists of four questions on pain in neck, back, and hip, morning stiffness, well-being, and pain/stiffness in other joints in addition to blood test of CRP. Score 0-4 (<1.3 inactive disease, >3,5 very high disease activity). Equation ASDAS-CRP = 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1)
Biomarker C-reaktivt protein (CRP) | after 3 months
  Venous blood to study CRP level by ELISA in µg/ml
Biomarker C-reaktivt protein (CRP) | after 12 months
  Venous blood to study CRP level by ELISA in µg/ml
Biomarker Pentraxin-related protein (PTX3) | after 3 months
  Venous blood to study PTX3 by ELISA in µg/ml
Biomarker Pentraxin-related protein (PTX3) | after 12 months
  Venous blood to study PTX3 by ELISA in µg/ml
Biomarker serum amyloid A1 | after 3 months
  Venous blood to study serum amyloid A1 by ELISA in µg/ml
Biomarker serum amyloid A1 | after 12 months
  Venous blood to study serum amyloid A1 by ELISA in µg/ml

SECONDARY OUTCOMES:
Aerobic capacity VO2max | after 3 months
  VO2max is measured according to Åstrand with a submaximal cycle ergometer test on an indoor stationary bicycle relative to body weight and expressed as the total amount of oxygen metabolized per minute per kilogram of body weight (mL/kg/min)
Aerobic capacity VO2max | after 12 months
  VO2max is measured according to Åstrand with a submaximal cycle ergometer test on an indoor stationary bicycle relative to body weight and expressed as the total amount of oxygen metabolized per minute per kilogram of body weight (mL/kg/min)
Blood pressure | after 3 months
  Blood pressure measured with an automatic blood pressure monitor (Omron M3, Omron Healthcare Co, Mukō, Japan) in millimetres of mercury (mmHg) and is giving numbers of systolic and diastolic pressures
Blood pressure | after 12 months
  Blood pressure measured with an automatic blood pressure monitor (Omron M3, Omron Healthcare Co, Mukō, Japan) in millimetres of mercury (mmHg) and is giving numbers of systolic and diastolic pressures
Grip strength | after 3 months
  The maximum hand grip strength (kg) measured with a hand dynamometer (KERN Sohn GmbH, Balingen, Germany) as another indicator of general body strength
Grip strength | after 12 months
  The maximum hand grip strength (kg) measured with a hand dynamometer (KERN Sohn GmbH, Balingen, Germany) as another indicator of general body strength
Body composition fat percent | after 3 months
  Proportion of fat % assessed by bioelectrical impedance analysis (Inbody 770®, Seoul, Korea)
Body composition fat percent | after 12 months
  Proportion of fat % assessed by bioelectrical impedance analysis (Inbody 770®, Seoul, Korea)
Body composition visceral fat area | after 3 months
  Proportion of visceral fat area assessed by bioelectrical impedance analysis (Inbody 770®, Seoul, Korea) in cm2 measures body adipose tissue without muscle, bone or other irrelevant structures
Body composition visceral fat area | after 12 months
  Proportion of visceral fat area assessed by bioelectrical impedance analysis (Inbody 770®, Seoul, Korea) in cm2 measures body adipose tissue without muscle, bone or other irrelevant structures
Body mass index (BMI) | after 3 months
  Measure based on kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
Body mass index (BMI) | after 12 months
  Measure based on kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
Self-reported physical function | after 3 months
  Measured with Bath Ankylosing Spondylitis Indices for function (BASFI) based on the mean of 10 questions with a total score 0-10 (best-worse)
Self-reported physical function | after 12 months
  Measured with Bath Ankylosing Spondylitis Indices for function (BASFI) based on the mean of 10 questions with a total score 0-10 (best-worse)
Self-reported Health status | after 3 months
  Measured with EuroQol-5 domain (EQ-5D) with five questions covering mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The total score range from 0-1 (no health to full health)
Self-reported Health status EuroQol-5 domain (EQ-5D) | after 12 months
  Measured with EuroQol-5 domain (EQ-5D) with five questions covering mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The total score range from 0-1 (no health to full health)
Self-reported well-being | after 3 months
  Measured with Assessment of SpondyloArthritis International Society Health Index (ASAS-HI) with 17 statements (yes/no) on pain, emotional functions, sleep, sexual functions, mobility, self-care and participation. Total score ranges from 0-17 (best-worse well-being)
Self-reported well-being | after 12 months
  Measured with Assessment of SpondyloArthritis International Society Health Index (ASAS-HI) with 17 statements (yes/no) on pain, emotional functions, sleep, sexual functions, mobility, self-care and participation. Total score ranges from 0-17 (best-worse well-being)
Self-reported pain | after 3 months
  Pain measured with a pain mannequin, with 18 predefined pain regions where participants mark their painful areas on the pain figure, total range 0-18
Self-reported pain | after 12 months
  Pain measured with a pain mannequin, with 18 predefined pain regions where participants mark their painful areas on the pain figure, total range 0-18
Self-reported pain intensity | after 3 months
  Pain intensity measured with numeric rating scale NRS 0-10, best to worst
Self-reported pain intensity | after 12 months
  Pain intensity measured with numeric rating scale NRS 0-10, best to worst
Self-reported Fatigue | after 3 months
  Measured with Fatigue Severity Scale (FSS). Consists of nine statements of the consequences of fatigue. The total score range from 9-63 (best-worst).
Self-reported Fatigue | after 12 months
  Measured with Fatigue Severity Scale (FSS). Consists of nine statements of the consequences of fatigue. The total score range from 9-63 (best-worst).
Objective adherence to physical activity and exercise recommendations | after 3 months
  Adherence to physical activity and exercise recommendations will be objectively measured through the heart rate monitor watch in average minutes of moderate/vigorous level of physical activity per week (of at least 75% of MHR).
Objective adherence to physical activity and exercise recommendations | after 12 months
  Adherence to physical activity and exercise recommendations will be objectively measured through the heart rate monitor watch in average minutes of moderate/vigorous level of physical activity per week (of at least 75% of MHR).
Self-reported adherence to physical activity and exercise recommendations | after 3 months
  Self-reported adherence to physical activity and exercise recommendations of at least 150 minutes of moderate-intensity aerobic physical activity throughout the week or doing at least 75 minutes of vigorous-intensity aerobic physical activity throughout the week or an equivalent combination of moderate - and vigorous-intensity activity (yes or no) will be collected through three validated questions including information on intensity, frequency, and duration
Self-reported adherence to physical activity and exercise recommendations | after 12 months
  Self-reported adherence to physical activity and exercise recommendations of at least 150 minutes of moderate-intensity aerobic physical activity throughout the week or doing at least 75 minutes of vigorous-intensity aerobic physical activity throughout the week or an equivalent combination of moderate - and vigorous-intensity activity (yes or no) will be collected through three validated questions including information on intensity, frequency, and duration
Self-reported confidence in one's own ability to manage pain | after 3 months
  Measured with the Arthritis Self-Efficacy Scale (ASES) for pain based on five questions with a total scores 10-100 (low to high self-efficacy).
Self-reported confidence in one's own ability to manage pain | after 12 months
  Measured with the Arthritis Self-Efficacy Scale (ASES) for pain based on five questions with a total scores 10-100 (low to high self-efficacy).
Self-reported confidence in one's own ability to manage symptoms | after 3 months
  Measured with the Arthritis Self-Efficacy Scale (ASES) for symptoms based on six questions with a total scores 10-100 (low to high self-efficacy).
Self-reported confidence in one's own ability to manage symptoms | after 12 months
  Measured with the Arthritis Self-Efficacy Scale (ASES) for symptoms based on six questions with a total scores 10-100 (low to high self-efficacy).
Self-reported confidence in one's own ability to do high-intensity exercise | after 3 months
  Measured with the Swedish Exercise Self-Efficacy Scale (S-ESES) based on 10 statements with the total score ranges from 10-40 (not at all safe to completely confident)
Self-reported confidence in one's own ability to do high-intensity exercise | after 12 months
  Measured with the Swedish Exercise Self-Efficacy Scale (S-ESES) based on 10 statements with the total score ranges from 10-40 (not at all safe to completely confident)
Proinflammatory cytokin TNF-α | after 3 months
  Venous blood to study serum TNF-α by Luminex in pg/ml
Proinflammatory cytokin TNF-α | after 12 months
  Venous blood to study serum TNF-α by Luminex in pg/ml
Proinflammatory cytokin IL-6 | after 3 months
  Venous blood to study serum IL-6 by Luminex in pg/ml
Proinflammatory cytokin IL-6 | after 12 months
  Venous blood to study serum IL-6 by Luminex in pg/ml
Proinflammatory cytokin IL-17a | after 3 months
  Venous blood to study serum IL-17a by Luminex in pg/ml
Proinflammatory cytokin IL-17a | after 12 months
  Venous blood to study serum IL-17a by Luminex in pg/ml
Proinflammatory cytokin IL-18 | after 3 months
  Venous blood to study serum IL-18 by Luminex in pg/ml
Proinflammatory cytokin IL-18 | after 12 months
  Venous blood to study serum IL-18 by Luminex in pg/ml
Proinflammatory cytokin IL-21 | after 3 months
  Venous blood to study serum IL-21 by Luminex in pg/ml
Proinflammatory cytokin IL-21 | after 12 months
  Venous blood to study serum IL-21 by Luminex in pg/ml
Proinflammatory cytokin IL-23 | after 3 months
  Venous blood to study serum IL-23 by Luminex in pg/ml
Proinflammatory cytokin IL-23 | after 12 months
  Venous blood to study serum IL-23 by Luminex in pg/ml
Chemokines CXCL10 | after 3 months
  Venous blood to study serum CXCL10, the Interferon gamma-induced protein 10 by Luminex in pg/ml
Chemokines CXCL10 | after 12 months
  Venous blood to study serum CXCL10, the Interferon gamma-induced protein 10 by Luminex in pg/ml
Inflammation-related protein Vascular endothelial growth factor (VEGF-A) | after 3 months
  Venous blood to study serum VEGF-A by Luminex in pg/ml
Inflammation-related protein Vascular endothelial growth factor (VEGF-A) | after 12 months
  Venous blood to study serum VEGF-A by Luminex in pg/ml
Inflammation-related protein interleukin 1 receptor antagonist (IL-1Ra) | after 3 months
  Venous blood to study serum IL-1Ra by Luminex in pg/ml
Inflammation-related protein interleukin 1 receptor antagonist (IL-1Ra) | after 12 months
  Venous blood to study serum IL-1Ra by Luminex in pg/ml
Inflammation-related protein Interleukin 8 (IL-8) | after 3 months
  Venous blood to study serum IL-8 by Luminex in pg/ml
Inflammation-related protein Interleukin 8 (IL-8) | after 12 months
  Venous blood to study serum IL-8 by Luminex in pg/ml
Inflammation-related protein Macrophage Inflammatory Proteins (MIP-1a) | after 3 months
  Venous blood to study serum MIP-1a by Luminex in pg/ml
Inflammation-related protein Macrophage Inflammatory Proteins (MIP-1a) | after 12 months
  Venous blood to study serum MIP-1a by Luminex in pg/ml
Inflammation-related protein macrophage inflammatory protein-1β (MIP-1β) | after 3 months
  Venous blood to study serum MIP-1β by Luminex in pg/ml
Inflammation-related protein macrophage inflammatory protein-1β (MIP-1β) | after 12 months
  Venous blood to study serum MIP-1β by Luminex in pg/ml
Protein serum calprotectin | after 3 months
  Venous blood to study serum calprotectin by ELISA in µg/ml
Protein serum calprotectin | after 12 months
  Venous blood to study serum calprotectin by ELISA in µg/ml
CRP/albumin ratio | after 3 months
  Venous blood to study serum CRP/albumin ratio by ELISA in mg/ml
CRP/albumin ratio | after 12 months
  Venous blood to study serum CRP/albumin ratio by ELISA in mg/ml
Myokine irisin | after 3 months
  Venous blood to study serum irisin by Luminex in ng/ml
Myokine irisin | after 12 months
  Venous blood to study serum irisin by Luminex in ng/ml
Myokine Brain-derived neurotrophic factor (BDNF) | after 3 months
  Venous blood to study serum BDNF by Luminex in ng/ml
Myokine Brain-derived neurotrophic factor (BDNF) | after 12 months
  Venous blood to study serum BDNF by Luminex in ng/ml
Bone and cartilage protein Dickkopf-related protein 1 (DKK-1) | after 3 months
  Venous blood to study serum DKK-1 by Luminex in pg/ml
Bone and cartilage protein Dickkopf-related protein 1 (DKK-1) | after 12 months
  Venous blood to study serum DKK-1 by Luminex in pg/ml
Bone and cartilage protein osteocalcin | after 3 months
  Venous blood to study serum osteocalcin by Luminex in ng/ml
Bone and cartilage protein osteocalcin | after 12 months
  Venous blood to study serum osteocalcin by Luminex in ng/ml
Bone and cartilage protein sclerostin | after 3 months
  Venous blood to study serum sclerostin by Luminex in ng/ml
Bone and cartilage protein sclerostin | after 12 months
  Venous blood to study serum sclerostin by Luminex in ng/ml
Bone and cartilage protein osteopontin | after 3 months
  Venous blood to study serum osteopontin by Luminex in ng/ml
Bone and cartilage protein osteopontin | after 12 months
  Venous blood to study serum osteopontin by Luminex in ng/ml
Bone and cartilage protein fibroblast growth factor 23 (FGF-23) | after 3 months
  Venous blood to study serum FGF-23 by Luminex in pg/ml
Bone and cartilage protein fibroblast growth factor 23 (FGF-23) | after 12 months
  Venous blood to study serum FGF-23 by Luminex in pg/ml
Bone and cartilage protein Bone morphogenetic protein 7 (BMP- 7) | after 3 months
  Venous blood to study serum BMP- 7 by Luminex in ng/ml
Bone and cartilage protein Bone morphogenetic protein 7 (BMP- 7) | after 12 months
  Venous blood to study serum BMP- 7 by Luminex in ng/ml
Bone and cartilage protein matrix metalloproteinase-3 (MMP-3) | after 3 months
  Venous blood to study serum MMP-3 by Luminex in ng/ml
Bone and cartilage protein matrix metalloproteinase-3 (MMP-3) | after 12 months
  Venous blood to study serum MMP-3 by Luminex in ng/ml
Liver-derived protein Fibroblast growth factor 21 (FGF-21) | after 3 months
  Venous blood to study serum FGF-21 by Luminex in ng/ml
Liver-derived protein Fibroblast growth factor 21 (FGF-21) | after 12 months
  Venous blood to study serum FGF-21 by Luminex in ng/ml
Apolipoprotein B (ApoB) | after 3 months
  Plasma samples to study lipoprotein ApoB will be sent to the hospital chemistry lab for current laboratory standards in g/L
Apolipoprotein B (ApoB) | after 12 months
  Plasma samples to study lipoprotein ApoB will be sent to the hospital chemistry lab for current laboratory standards in g/L
Apolipoprotein A1 (ApoA1) | after 3 months
  Plasma samples to study lipoprotein ApoA1 will be sent to the hospital chemistry lab for current laboratory standards in g/L
Apolipoprotein A1 (ApoA1) | after 12 months
  Plasma samples to study lipoprotein ApoA1 will be sent to the hospital chemistry lab for current laboratory standards in g/L

CONTACTS AND LOCATIONS:
Overall Officials: Haglund, Assoc. prof., Principal Investigator — Dept. of Environmental and Biosciences, Halmstad University, Sweden
Locations (1):
- Halmstad University, Halmstad, Halland County, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT05781763/Prot_SAP_000.pdf